CLINICAL TRIAL: NCT01824082
Title: Treating Intractable Post-Amputation Phantom Limb Pain With Ambulatory Continuous Peripheral Nerve Blocks
Brief Title: Treating Phantom Limb Pain Using Continuous Peripheral Nerve Blocks: A Department of Defense Funded Multicenter Study
Acronym: DoD-PLP-Tx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phantom Pain Treatment (DoD)
Record Dates: First submitted 2013-03-30; First posted 2013-04-04 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Phantom Limb Pain
Keywords: phantom pain; traumatic limb amputation; amputees
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators originally planned to unmask the treatment groups following the completion of the statistical analysis ("triple masked"); but following the analysis using "treatment A" and "treatment B" labels, opted to wait to unmask the groups until the manuscript was drafted ("quadruple masking").
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine 0.5% (Experimental): Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of study fluid from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. Subjects assigned this treatment for their initial infusion will have the option of returning 4-16 weeks later for a second infusion of the alternate treatment: normal saline.
  Interventions: Drug: Perineural infusion [continuous peripheral nerve block(s)]
- Normal saline (salt water) infusion (Placebo Comparator): Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of normal saline placebo fluid from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. Subjects assigned this treatment for their initial infusion will have the option of returning 4-16 weeks later for a second infusion of the alternate treatment: ropivacaine 0.5%.
  Interventions: Drug: Perineural infusion [continuous peripheral nerve block(s)]

INTERVENTIONS:
Drug: Perineural infusion [continuous peripheral nerve block(s)] — Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of study fluid from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. Subjects will have the option of returning 4-16 weeks later for a second infusion of the alternate treatment solution.

SUMMARY:
When a limb is traumatically severed, pain perceived in the part of the body that no longer exists often develops. This is called "phantom limb" pain, and is different from "stump" pain, which is pain within the part of the limb that remains intact. Unfortunately, phantom pain resolves in only 16% of people, with the rest experiencing this pain for the remainder of the lives. There is currently no reliable treatment for phantom limb pain.

The exact reason that phantom limb pain occurs is unclear, but when a nerve is cut-as happens with a traumatic amputation-changes occur in the brain and spinal cord that actually worsen with increasing phantom pain. These abnormal changes may often be corrected by putting local anesthetic-termed a "peripheral nerve block"-on the injured nerve, keeping any "bad signals" from reaching the brain, with resolution of the phantom limb pain. However, when the nerve block ends after a few hours, the phantom pain returns. But, this demonstrates that the brain abnormalities-and phantom pain-that occur with an amputation may be dependent upon the "bad" signals being sent from the injured nerve(s), suggesting that a very long peripheral nerve block-lasting many days rather than hours-may permanently reverse the abnormal changes in the brain, and provide lasting relief from phantom pain.

Until recently, extending a peripheral nerve block beyond 16 hours was unrealistic. However, a treatment option called a "continuous peripheral nerve block" is now available. This technique involves the placement of a tiny tube-smaller than a piece of spaghetti-through the skin and next to the nerves supplying the amputated limb. The tiny tube may be placed with minimal discomfort in about 15 minutes. Numbing medicine called local anesthetic is then infused through the tube, blocking any signals that the injured nerve sends to the spinal cord and brain. Using a small, portable infusion pump, this prolonged nerve block may be provided in individuals' own homes.

The ultimate objective of the proposed research study is to determine if a 6-day continuous peripheral nerve block provided at home is an effective treatment for persistent phantom limb pain following a traumatic limb amputation. The primary hypothesis (what the researchers predict) is that phantom limb pain intensity will be significantly decreased 4 weeks following treatment with a 6-day continuous peripheral nerve block.

DETAILED DESCRIPTION:
Background. The combination of increased munitions force, use of improvised explosive devices, and casualty survival rates has resulted in a dramatic increase in the percentage of injured combat veterans living with a traumatic amputation. Of American Veteran amputees, 35-98% develop chronic, intractable pain perceived as being from the missing limb, a phenomenon termed "phantom limb pain." This pain resolves in only 16% of afflicted individuals, and there is currently no reliable treatment. The etiology of phantom pain remains unclear, but evidence suggests that severing a nerve provokes changes in the spinal cord, thalamus, and cerebral cortex. When neural input from an amputated limb is blocked with local anesthetic (a peripheral nerve block), cortical abnormalities and phantom pain frequently resolve. However, when the single-injection nerve block resolves after a few hours, the phantom pain returns. These findings demonstrate that cortical abnormalities and phantom pain may be maintained from abnormal peripheral input, suggesting that a peripheral nerve block of extended duration-lasting many days rather than hours-may permanently reorganize cortical pain mapping, thus providing lasting relief from phantom pain. A "continuous peripheral nerve block" (CPNB) involves the percutaneous insertion of a catheter directly adjacent to the peripheral nerves supplying an affected limb. Local anesthetic infused via the catheter(s) induces a completely insensate extremity for as long as desired without any systemic side effects. Additionally, CPNB may be provided on an ambulatory basis using a small, portable pump to infuse the local anesthetic.

Objective. To determine if ambulatory CPNB is an effective treatment for intractable phantom limb pain following a traumatic limb amputation. Previously-published small, uncontrolled series describe patients immediately following surgical amputation whose phantom limb pain dramatically decreased or completely resolved with CPNB. We have data from a randomized, double-masked, placebo-controlled, crossover pilot study suggesting great promise treating intractable phantom limb pain with ambulatory CPNB: participants (n=3) experienced no change in their phantom pain following a 6-day infusion of normal saline; however, with a 6-day CPNB of potent local anesthetic administered 4 months later, subjects (n=2; one patient returned to duty before crossover infusion) experienced complete resolution of their phantom limb pain. Within the 12-week follow-up period, one subject experienced no phantom pain recurrence; and the other subject reported mild pain occurring once each week of just a small fraction of his original pain.

Specific Aims. The primary hypothesis is that phantom limb pain intensity will be significantly decreased 4 weeks following an ambulatory CPNB (as measured by the Numeric Rating Scale of the Brief Pain Inventory).

Study Design. We propose a multicenter, randomized, double-masked, placebo-controlled, simultaneous parallel and crossover, human-subjects clinical trial. We will include subjects with an existing upper or lower amputation who experience phantom limb pain at least daily for the previous 4 weeks. Catheter site(s) will be determined by amputation location. Subjects will be randomized to receive one of two study solutions in a double-masked manner: either a local anesthetic (ropivacaine 0.5%) or placebo (normal saline). Catheters will be removed after 6 days of at-home infusion. Although not required, each subject has the option to return for the alternative treatment four weeks later (crossover infusion). The primary endpoint will be the difference in average phantom pain intensity at baseline and 4 weeks following the initial infusion as measured with the Numeric Rating Scale between treatment groups for the initial infusion. Major secondary endpoints will involve intra- and inter-subject comparisons of additional measures of pain and health-related quality-of-life.

Clinical Impact. From 2001-2006, over 70% of all U.S. military casualties endured a major limb injury, with an amputation rate of 28% within Operation Enduring Freedom alone. Previous conflicts have left tens-of-thousands of United States Armed Forces Veterans with missing limbs. CPNB are now relatively ubiquitous within the United States, but applied nearly exclusively to provide acute post-injury/surgical analgesia. If the proposed study demonstrates that ambulatory CPNB is a reliable treatment for intractable phantom limb pain, the resulting impact in treating the consequences of traumatic amputation will be immediate and profound, as healthcare providers within the United States Armed Forces and Veterans Affairs Medical Centers already have expertise placing and managing perineural catheters. Currently, CPNB is provided exclusively in the acute setting-to treat pain immediately following a battlefield injury or surgery-and not chronic, intractable phantom limb pain. However, because there is little technical difference in providing CPNB for acute versus chronic pain, the thousands of U.S. Veterans and active duty personnel suffering from intractable phantom pain could be treated relatively easily, rapidly, and with negligible additional costs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Upper or lower limb traumatic or surgical amputation at least 12 weeks prior to enrollment at or distal to the mid-humerus or hip (femoral head remaining), respectively; and including at least one metacarpal or metatarsal bone, respectively.
* Experiencing at least moderate phantom limb pain (defined as 2 or higher on the numeric rating scale, NRS 0-10), at least three times each week for the previous 8 weeks.
* Accepting of an ambulatory continuous peripheral nerve block for 6 days.
* Willing to avoid changes to their analgesic regimen from 4 weeks prior to and at least 4 weeks following the initial catheter placement (preferably 4 weeks following the second/crossover catheter insertion as well).
* Having a "caretaker" who will transport the subject home following the catheter insertion(s), and remain with the subject for the first night of the infusions.

Exclusion Criteria:

* Known renal insufficiency
* Allergy to study medications
* Pregnancy
* Incarceration
* Inability to communicate with the investigators
* Morbid obesity (BMI greater than 40)
* Comorbidity that results in moderate-to-severe functional limitation (ASA greater than 2)
* Possessing any contraindication to ambulatory perineural catheter placement or perineural local anesthetic infusion:

  * Current infection
  * Immune-compromised status of any etiology
  * Uncontrolled anxiety/panic disorder
  * Inability to contact investigators during the perineural infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - Veteran's Affairs Palo Alto Health Care System, Palo Alto, California
  - University of California, San Diego, Hillcrest Medical Center, San Diego, California
  - Walter Reed Army National Medical Center, Bethesda, Maryland
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Ilfeld BM, Khatibi B, Maheshwari K, Madison S, Ali Sakr Esa W, Mariano ER, Kent M, Hanling S, Sessler DI, Eisenach JC, Cohen SP, Mascha E, Li S, Turan A; PAINfRE Investigators. Patient-centered results from a multicenter study of continuous peripheral nerve blocks and postamputation phantom and residual limb pain: secondary outcomes from a randomized, clinical trial. Reg Anesth Pain Med. 2023 Sep;48(9):471-477. doi: 10.1136/rapm-2023-104389. Epub 2023 Mar 9. PMID 36894197
- [Derived] Ilfeld BM, Khatibi B, Maheshwari K, Madison SJ, Ali Sakr Esa W, Mariano ER, Kent ML, Hanling S, Sessler DI, Eisenach JC, Cohen SP, Mascha EJ, Yang D, Padwal JA, Turan A; PAINfRE Investigators. Immediate Effects of a Continuous Peripheral Nerve Block on Postamputation Phantom and Residual Limb Pain: Secondary Outcomes From a Multicenter Randomized Controlled Clinical Trial. Anesth Analg. 2021 Oct 1;133(4):1019-1027. doi: 10.1213/ANE.0000000000005673. PMID 34314392
- [Derived] Ilfeld BM, Khatibi B, Maheshwari K, Madison SJ, Esa WAS, Mariano ER, Kent ML, Hanling S, Sessler DI, Eisenach JC, Cohen SP, Mascha EJ, Ma C, Padwal JA, Turan A; PAINfRE Investigators. Ambulatory continuous peripheral nerve blocks to treat postamputation phantom limb pain: a multicenter, randomized, quadruple-masked, placebo-controlled clinical trial. Pain. 2021 Mar 1;162(3):938-955. doi: 10.1097/j.pain.0000000000002087. PMID 33021563

RESULTS

PARTICIPANT FLOW:
Period: Initial Treatment
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Started | 71 | 73
Completed | 71 | 73
Not Completed | 0 | 0
Period: Optional Crossover Treatment
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Started | 40 | 25
Completed | 40 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 73 | 144
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 30 | 51
  Male | 50 | 43 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 71 | 73 | 144
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27 [25 to 31] | 27 [24 to 33] | 27 [24 to 32]
Marital status [Count of Participants; unit: Participants]
  Single (or divorced) | 31 | 37 | 68
  Currently married | 37 | 26 | 63
  Others (separated and widowed) | 3 | 10 | 13
Military Status [Count of Participants; unit: Participants]
  Civilian (never in military) | 56 | 61 | 117
  Veteran | 14 | 12 | 26
  Active Duty | 1 | 0 | 1
Years of education [Median (Inter-Quartile Range); unit: years] | 14 [12 to 16] | 13 [12 to 16] | 13 [12 to 16]
Amputation Information [Count of Participants; unit: Participants]
  Lower extremity above knee | 28 | 24 | 52
  Lower extremity below knee | 30 | 39 | 69
  Upper extremity above elbow | 11 | 8 | 19
  Upper extremity below elbow | 2 | 2 | 4
  Right (vs. left) side | 32 | 37 | 69
  Traumatic amputation | 20 | 16 | 36
  Surgical amputation due to cancer | 5 | 5 | 10
  Surgical amputation due to infection | 27 | 32 | 59
  Surgical amputation due to trauma | 7 | 6 | 13
  Surgical amputation due to vascular deficiency | 8 | 8 | 16
  Surgical amputation due to other cause | 4 | 6 | 10
  History of residual limb pain | 50 | 57 | 107
  Current residual limb pain | 40 | 48 | 88
  Current prosthesis use | 50 | 60 | 110
  Additional limb amputation(s) | 12 | 11 | 23
Pain immediately before and after initial local anesthetic bolus measured on the 0-10 NRS [Median (Inter-Quartile Range); unit: units on a scale] — Measured by the Numeric Rating Scale . The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, with zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
  units on a scale
    Phantom pain immediately before bolus | 5 [3 to 7] | 5 [3 to 7] | 5 [3 to 7]
    Phantom pain 20 minutes after bolus | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
    Residual limb pain immediately before bolus | 1 [0 to 4] | 3 [0 to 5] | 2 [0 to 5]
    Residual limb pain 20 minutes after bolus | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Phantom Pain previous 3 days as measured on the 0-10 NRS [Median (Inter-Quartile Range); unit: units on a scale] — Measured by the Numeric Rating Scale Within the Brief Pain Inventory. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, with zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
  units on a scale
    Current | 5.0 [2.0 to 7.0] | 5.0 [3.0 to 7.0] | 5.0 [2.0 to 7.0]
    Least | 2.0 [1.0 to 4.0] | 3.0 [2.0 to 5.0] | 2.0 [1.0 to 5.0]
    Average | 5.0 [4.0 to 7.0] | 5.0 [4.0 to 7.0] | 5.0 [4.0 to 7.0]
    Worst | 8.0 [8.0 to 10.0] | 8.0 [7.0 to 10.0] | 8.0 [7.0 to 10.0]
Residual limb pain previous 3 days ( Numeric Rating Scale) [Median (Inter-Quartile Range); unit: units on a scale] — Measured by the Numeric Rating Scale Within the Brief Pain Inventory. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, with zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
  units on a scale
    Current | 1.0 [0 to 4.0] | 3.0 [0 to 6.0] | 2.0 [0 to 5.0]
    Least | 0 [0 to 3.0] | 2 [0 to 4.0] | 1 [0 to 4]
    Average | 3 [0 to 5.0] | 4.0 [1.0 to 6.0] | 3 [0 to 6]
    Worst | 5 [0 to 8.0] | 6.0 [2.0 to 8.0] | 5 [0 to 8]
Phantom pain relief from medication (%) [Count of Participants; unit: Participants] — Measured as part of the Brief Pain inventory: the percentage of phantom limb pain that is relieved when medication is taken
  Participants
    0-25% | 26 | 22 | 48
    26-50% | 21 | 18 | 39
    51-75% | 5 | 13 | 18
    76-100% | 8 | 4 | 12
    Did not use any medication or pain treatment | 11 | 16 | 27
Residual pain relief from medication (%) [Count of Participants; unit: Participants] — Measured as part of the Brief Pain inventory: the percentage of residual limb pain that is relieved when medication is taken
  Participants
    0-25% | 23 | 19 | 42
    26-50% | 10 | 16 | 26
    51-75% | 5 | 9 | 14
    76-100% | 8 | 3 | 11
    Did not use any medication or pain treatment | 25 | 26 | 51
Pain Interference components ( Brief Pain Inventory) [Median (Inter-Quartile Range); unit: units on a scale] — The Brief Pain Inventory is an instrument that includes-in addition to pain intensity scales-seven measures evaluating pain's interference with physical and emotional functioning, such as sleep, relations with others, and enjoyment of life. Measured in a scale of 0-10, where 0=does not interfere, 10=Completely interferes.
  units on a scale
    General activity | 6.0 [3.0 to 8.0] | 5.0 [3.0 to 8.0] | 5 [3 to 8]
    Mood | 6.0 [2.0 to 9.0] | 6.0 [4.0 to 8.0] | 6 [3 to 9]
    Walking ability | 5.0 [0 to 9.0] | 5.0 [2.0 to 9.0] | 5 [0 to 9]
    Normal work | 6.0 [3.0 to 8.0] | 5.0 [2.0 to 8.0] | 5 [2 to 8]
    Relations with other people | 4.0 [0 to 7.0] | 4.0 [0 to 7.0] | 4 [0 to 7]
    Sleep | 8.0 [5.0 to 9.0] | 7.0 [4.0 to 8.0] | 7 [4 to 9]
    Enjoyment of life | 6.0 [2.0 to 9.0] | 6.0 [3.0 to 8.0] | 6 [2 to 9]
Depression as measured with the Beck's Depression Inventory [Median (Inter-Quartile Range); unit: units on a scale] — The Beck Depression Inventory is a 21-item instrument that measures characteristic symptoms and signs of depression, requires only a 5th grade comprehension level to adequately understand the questions, and demonstrates a high internal consistency (0.73-0.92, mean of 0.86), reliability and validity. Each of the 21 factors is rated on a 0-3 scale, and then summed to produce the total score of 0-63. Mild, moderate, and severe depression is defined with scores of 10-18, 19-29, and 30-63, respectively.
  units on a scale | 15 [4 to 24] | 14 [7 to 24] | 14 [4 to 24]
Beck Depression Inventory [Count of Participants; unit: Participants] — The Beck Depression Inventory is a 21-item instrument measuring characteristic symptoms and signs of depression. Each of the 21 factors is rated on a 0-3 scale, and then summed to produce the total score of 0-63. Mild, moderate, and severe depression are defined with scores of 10-18, 19-29, and 30-63, respectively.
  Participants
    Minimal depression | 25 | 30 | 55
    Mild depression | 16 | 14 | 30
    Moderate depression | 24 | 20 | 44
    Severe depression | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: "Average" Phantom Limb Pain Intensity 4 Weeks Following Initiation of an Ambulatory Continuous Peripheral Nerve Block (as Measured by the Numeric Rating Scale Within the Brief Pain Inventory)
Description: Phantom pain will be assessed using a Numeric Rating Scale (NRS) as part of the Brief Pain Inventory (short form), with the "average" pain score designated as the primary endpoint. In addition, average and worst residual limb pain NRS will be recorded separately from the phantom pain scores. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, with zero equivalent to no pain and 10 equivalent to the worst imaginable pain. These data are 4 weeks after the initiation of the FIRST intervention (and not the optional crossover treatment).
Time Frame: 4 weeks following the initiation of the initial intervention.
Population: "Average Phantom Limb Pain Intensity" at 4 weeks following the initiation of the first intervention before participants had the option to crossover to the other intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale | 3.0 (2.9) | 4.5 (2.6)

2. Secondary Outcome: Perception of Well-being (as Measured With the Patient Global Impression of Change Scale).
Description: The Patient Global Impression of Change Scale is a 7-point ordinal scale requiring the subject to rate the current severity of their global situation as it relates to phantom limb pain (as defined by each individual) compared to their baseline. This scale has the words "very much worse" to the left by the number one, and "very much improved" to the right, adjacent to the number seven. The words "no change" are in the middle of the scale above the number four. The Patient Global Impression of Change Scale has been validated in over ten prospective trials, including studies specifically involving peripheral neuropathy. These data are from 4 weeks after the initiation of the FIRST intervention (and not the optional crossover treatment).
Time Frame: 4 weeks following the initiation of the initial intervention
Population: Perception of well-being(as measured with the Patient Global Impression of Change Scale) at 4 weeks following the initiation of the first intervention before participants had the option to crossover to the other intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale | 5.0 [4.0 to 7.0] | 4.0 [4.0 to 5.0]

3. Secondary Outcome: Physical and Emotional Functioning 4 Weeks Following Initiation of Intervention (as Measured With the Brief Pain Inventory Interference Domain).
Description: The Brief Pain Inventory (interference sub scale) is an instrument that measures the interference with physical and emotional functioning using a 0-10 scale (0 = no interference; 10 = complete interference). The seven interference questions involve general activity, mood, walking ability, normal work activities (both inside and outside of the home), relationships, sleep, and enjoyment of life. The seven functioning questions can be added to produce an interference subscale (0-70). The use of both single items (e.g., mood) and the composite scores is supported. These data are from 4 weeks after the initiation of the FIRST intervention (and not the optional crossover treatment).
Time Frame: 4 weeks following initiation of the initial intervention
Population: Physical and emotional functioning ( as measured with the Brief Pain Inventory Interference Domain) at 4 weeks following the initiation of the first intervention before participants had the option to crossover to the other intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Total of 7 components | 11 [0 to 38] | 28 [4 to 45]
  General activity | 1.0 [0 to 6.0] | 5.0 [0 to 7.0]
  Mood | 0 [0 to 6.0] | 5.0 [0 to 8.0]
  Walking ability | 0 [0 to 3.0] | 3.0 [0 to 7.0]
  Normal Work | 0 [0 to 6.0] | 3.0 [0 to 6.0]
  Relations with others | 0 [0 to 5.0] | 2.5 [0 to 6.5]
  Sleep | 2.5 [0 to 8.0] | 5.5 [0 to 8.0]
  Enjoyment of life | 1.0 [0 to 7.0] | 4.0 [0 to 7.0]

4. Secondary Outcome: Depression 4 Weeks Following Initiation of Intervention (as Measured With the Beck Depression Inventory).
Description: The Beck Depression Inventory is a 21-item instrument that measures characteristic symptoms and signs of depression, requires only a 5th grade comprehension level to adequately understand the questions, and demonstrates a high internal consistency (0.73-0.92, mean of 0.86), reliability and validity. Each of the 21 factors is rated on a 0-3 scale, and then summed to produce the total score of 0-63. Mild, moderate, and severe depression is defined with scores of 10-18, 19-29, and 30-63, respectively. This data is 4 weeks following the initiation of the initial intervention, and NOT the optional crossover treatment.
Time Frame: 4 weeks following initiation of the initial intervention
Population: Depression(as measured with the Beck Depression Inventory) at 4 weeks following the initiation of the first intervention before participants had the option to crossover to the other intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale | 6 [2 to 17] | 13 [4 to 22]

5. Other Pre Specified Outcome: Change in Physical and Emotional Functioning at 6 and 12 Months Compared With Baseline (as Measured With the Brief Pain Inventory Interference Domain).
Description: The Brief Pain Inventory (interference sub scale) is an instrument that measures the interference with physical and emotional functioning using a 0-10 scale (0 = no interference; 10 = complete interference). The seven interference questions involve general activity, mood, walking ability, normal work activities (both inside and outside of the home), relationships, sleep, and enjoyment of life. The seven functioning questions can be added to produce an interference subscale (0-70). The use of both single items (e.g., mood) and the composite scores is supported. The reported data is the reported interference sub scale at 6 and 12 months compared with baseline.
Time Frame: 6 and 12 months following initiation of the initial intervention
Population: All subjects received the initial intervention. However, only a subset of each group chose to participate in the optional crossover treatment that occurred 1-4 months following the initiation of the initial treatment infusion. For those who did participate in the optional crossover treatment, they received the alternative treatment as their initial treatment (e.g., subjects who initially received placebo saline subsequently received Ropivacaine 0.5%, and vice versa).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Ropivacaine 0.5% Only (no Placebo Crossover): Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of ropivacaine 0.5% from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. Subjects assigned this treatment for their initial infusion will have the option of returning 4-16 weeks later for a second infusion of the alternate treatment: normal saline.
- Placebo Infusion Only (no Ropivacaine 0.5% Crossover): Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of normal saline placebo fluid from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. Subjects assigned this treatment for their initial infusion will have the option of returning 4-16 weeks later for a second infusion of the alternate treatment: ropivacaine 0.5%.
- Ropivacaine 0.5% Followed by Placebo Infusion: Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of ropivacaine 0.5% from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). Subjects assigned this treatment returned 4-16 weeks later for a second infusion of the alternate treatment: normal saline.
- Placebo Followed by Ropivacaine 0.5% Infusion: Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of normal saline placebo fluid from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. Subjects in this group returned returned 4-16 weeks later for a second infusion of the alternate treatment: ropivacaine 0.5%.
Arm/Group | Ropivacaine 0.5% Only (no Placebo Crossover) | Placebo Infusion Only (no Ropivacaine 0.5% Crossover) | Ropivacaine 0.5% Followed by Placebo Infusion | Placebo Followed by Ropivacaine 0.5% Infusion
Number analyzed (Participants) | 46 | 33 | 25 | 40
score on a scale
  General activity (6months following initiation of intervention) | -1.5 [-6.0 to 0] | -2.0 [-5.0 to 1.0] | 0 [-1.5 to 1.0] | -2.0 [-5.0 to 0]
  Mood (6months following initiation of intervention) | -1.0 [-5.0 to 0] | -1.0 [-4.0 to 0] | 0 [-2.0 to 1.0] | -1.0 [-5.0 to 0]
  Walking ability (6months following initiation of intervention) | 0 [-7.0 to 0] | -1.0 [-5.0 to 0] | 0 [-1.0 to 0] | -1.0 [-3.0 to 0]
  Normal work (6months following initiation of intervention) | -2.5 [-6.5 to 0] | -1.0 [-5.0 to 0] | 0 [-1.5 to 1.0] | -1.0 [-6.0 to 0]
  Relations with others (6months following initiation of intervention) | -1.0 [-5.5 to 0] | 0 [-5.0 to 0] | 0 [-1.5 to 1.0] | 0 [-3.0 to 1.0]
  Sleep (6months following initiation of intervention) | -3.8 [-7.0 to 0] | -1.5 [-6.0 to 0] | 0 [-1.00 to 0] | 0 [-6.0 to 0]
  Enjoyment of life (6months following initiation of intervention) | -2.0 [-7.5 to 0] | -1.0 [-5.0 to 0] | 0 [-2.0 to 0] | -2.0 [-5.0 to 0]
  General activity (12 months following initiation of intervention) | -1.0 [-4.0 to 0] | -1.0 [-5.0 to 0] | -1.0 [-4.0 to 1.0] | -1.0 [-3.5 to 0]
  Mood (12 months following initiation of intervention) | 0 [-4.0 to 0] | -1.0 [-4.0 to 0] | -1.0 [-4.0 to 0] | -0.5 [-3.8 to 1.0]
  Walking ability (12 months following initiation of intervention) | -1.0 [-6.0 to 0] | 0 [-5.0 to 0] | 0 [-3.0 to 0] | 0 [-4.5 to 0]
  Normal work (12 months following initiation of intervention) | -1.0 [-5.0 to 0] | -1.0 [-5.0 to 0] | -3.0 [-6.0 to 0] | -1.5 [-5.3 to 0]
  Relations with others (12 months following initiation of intervention) | -1.0 [-2.0 to 0] | 0 [-3.0 to 0] | -1.0 [-4.0 to 0] | -0.5 [-4.0 to 1.0]
  Sleep (12 months following initiation of intervention) | -1.0 [-6.0 to 0] | 0 [-6.0 to 0] | -1.0 [-2.0 to 0] | -0.5 [-6.5 to 0.5]
  Enjoyment of life (12 months following initiation of intervention) | -1.0 [-5.0 to 0] | -1.0 [-6.0 to 1.0] | 0 [-5.0 to 0] | 0 [-3.5 to 1.0]

6. Other Pre Specified Outcome: Change in Depression 6 and 12 Months Compared With Baseline (as Measured With the Beck Depression Inventory).
Description: The Beck Depression Inventory is a 21-item instrument that measures characteristic symptoms and signs of depression, requires only a 5th grade comprehension level to adequately understand the questions, and demonstrates a high internal consistency (0.73-0.92, mean of 0.86), reliability and validity. Each of the 21 factors is rated on a 0-3 scale, and then summed to produce the total score of 0-63. Mild, moderate, and severe depression is defined with scores of 10-18, 19-29, and 30-63, respectively. The data presented are the Beck Depression Inventory at 6 and 12 months compared with baseline.
Time Frame: 6 and 12 months following initiation of the initial intervention
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine 0.5% Only (no Placebo Crossover) | Placebo Infusion Only (no Ropivacaine 0.5% Crossover) | Ropivacaine 0.5% Followed by Placebo Infusion | Placebo Followed by Ropivacaine 0.5% Infusion
Number analyzed (Participants) | 46 | 33 | 25 | 40
units on a scale
  Month 6 | -3.0 [-11.0 to 0] | -2.0 [-6.0 to 0] | -1.5 [-2.0 to 0] | -4.0 [-8.0 to 0]
  Month 12 | -4.0 [-12.0 to -1.0] | -2.0 [-9.0 to 0] | -1.5 [-3.0 to 0] | -4.0 [-9.0 to -1.0]

7. Other Pre Specified Outcome: Perception of Well-being (as Measured With the Patient Global Impression of Change Scale).
Description: The Patient Global Impression of Change Scale is a 7-point ordinal scale requiring the subject to rate the current severity of their global situation as it relates to phantom limb pain (as defined by each individual) compared to their baseline. This scale has the words "very much worse" to the left by the number one, and "very much improved" to the right, adjacent to the number seven. The words "no change" are in the middle of the scale above the number four. The Patient Global Impression of Change Scale has been validated in over ten prospective trials, including studies specifically involving peripheral neuropathy.
Time Frame: 6 and 12 months following initiation of intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine 0.5% Only (no Placebo Crossover) | Placebo Infusion Only (no Ropivacaine 0.5% Crossover) | Ropivacaine 0.5% Followed by Placebo Infusion | Placebo Followed by Ropivacaine 0.5% Infusion
Number analyzed (Participants) | 46 | 33 | 25 | 40
units on a scale
  6 months following initiation of intervention | 7.0 [4.0 to 7.0] | 5.0 [4.0 to 7.0] | 4.0 [4.0 to 5.0] | 4.0 [4.0 to 7.0]
  12 months following initiation of intervention | 6.0 [4.0 to 7.0] | 5.0 [4.0 to 7.0] | 4.0 [4.0 to 7.0] | 4.0 [4.0 to 7.0]

8. Other Pre Specified Outcome: Masking Assessment
Description: Subjects were asked which study fluid they believed they were receiving during the initial infusion: The possible responses were:
  ☐Definitely active ☐Probably active ☐Does not know ☐ Probably saline ☐ Definitely saline
Time Frame: 4 weeks following the initial intervention
Population: Data analysed 28 days following the initial intervention and before the crossover treatment. So its analysed based on participants included in each arm group for the initial treatment. Not applicable for crossover treatment option.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
Participants
  Definitely Active | 10 | 2
  Probably Active | 17 | 8
  Does not know | 18 | 18
  Probably Saline | 16 | 33
  Definitely Saline | 3 | 4
  Missing | 7 | 8

9. Other Pre Specified Outcome: "Average" Phantom Limb Pain
Description: The "average" phantom limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21
Population: Days 1, 7, 14, 21 following the initiation of the first intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0 [0 to 2.5] | 3.3 [0 to 5.0]
  Day 7 | 2.0 [0 to 5.0] | 4.0 [0 to 5.0]
  Day 14 | 3.0 [0 to 6.0] | 4.5 [0 to 6.0]
  Day 21 | 3.0 [0 to 5.0] | 4.0 [0 to 6.0]

10. Other Pre Specified Outcome: "Worst" Phantom Limb Pain
Description: The worst phantom limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21, 28
Population: Days 1, 7, 14, 21 and 28 following the initiation of the first intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0.50 [0 to 5.0] | 5.0 [0 to 8.0]
  Day 7 | 4.0 [0.00 to 8.0] | 7.0 [2.5 to 8.3]
  Day 14 | 6.8 [1.00 to 8.5] | 7.0 [3.5 to 10.0]
  Day 21 | 5.0 [1.00 to 8.0] | 7.0 [4.0 to 9.0]
  Day 28 | 5.0 [1.00 to 8.0] | 8.0 [5.5 to 9.0]

11. Other Pre Specified Outcome: "Least" Phantom Limb Pain
Description: The least phantom limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21, 28.
Population: Days 1, 7, 14, 21 and 28 following the initiation of the first intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0 [0 to 0] | 0 [0 to 3.0]
  Day 7 | 0 [0 to 3.0] | 1.3 [0 to 3.0]
  Day 14 | 1.0 [0 to 4.5] | 1.0 [0 to 4.0]
  Day 21 | 1.0 [0 to 3.0] | 1.5 [0 to 5.0]
  Day 28 | 0 [0 to 3.0] | 2.0 [0 to 4.0]

12. Other Pre Specified Outcome: "Current" Phantom Limb Pain
Description: The current phantom limb pain at the time of the data collection phone call evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21, 28.
Population: Days 1, 7, 14, 21 and 28 following the initiation of the first intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0 [0 to 2.0] | 3.0 [0 to 6.0]
  Day 7 | 0 [0 to 5.0] | 3.0 [0 to 6.0]
  Day 14 | 2.0 [0 to 5.5] | 4.0 [0 to 6.0]
  Day 21 | 1.00 [0 to 5.0] | 4.0 [0 to 6.0]
  Day 28 | 0.50 [0 to 4.0] | 4.0 [0 to 7.0]

13. Other Pre Specified Outcome: "Average" Residual Limb Pain
Description: The "average" residual limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21, 28
Population: Days 1, 7, 14, 21 and 28 following the initiation of the first intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0 [0 to 0] | 0 [0 to 4.3]
  Day 7 | 0 [0 to 2.0] | 1.0 [0 to 4.0]
  Day 14 | 0 [0 to 3.0] | 1.5 [0 to 5.0]
  Day 21 | 0 [0 to 4.0] | 1.0 [0 to 5.0]
  Day 28 | 0 [0 to 2.5] | 3.0 [0 to 5.0]

14. Other Pre Specified Outcome: "Worst" Residual Limb Pain
Description: The worst residual limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21, 28.
Population: Days 1, 7, 14, 21 and 28 following the initiation of the first intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0 [0 to 0] | 0.50 [0 to 6.0]
  Day 7 | 0 [0 to 3.0] | 3.0 [0 to 6.0]
  Day 14 | 0 [0 to 7.0] | 4.0 [0 to 7.0]
  Day 21 | 0 [0 to 7.0] | 4.0 [0 to 7.0]
  Day 28 | 0 [0 to 5.0] | 6.0 [0 to 8.0]

15. Other Pre Specified Outcome: "Least" Residual Limb Pain
Description: The least residual limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21, 28
Population: Days 1, 7, 14, 21 and 28 following the initiation of the first intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0 [0 to 0] | 0 [0 to 4.3]
  Day 7 | 0 [0 to 2.0] | 1.0 [0 to 4.0]
  Day 14 | 0 [0 to 3.0] | 1.5 [0 to 5.0]
  Day 21 | 0 [0 to 4.0] | 1.0 [0 to 5.0]
  Day 28 | 0 [0 to 2.5] | 3.0 [0 to 5.0]

16. Other Pre Specified Outcome: "Current" Residual Limb Pain
Description: The current residual limb pain at the time of the data collection phone call evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Days 1, 7, 14, 21, 28.
Population: Days 1, 7, 14, 21 and 28 following the initiation of the first intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1 | 0 [0 to 0] | 0 [0 to 4.0]
  Day 7 | 0 [0 to 1.0] | 0 [0 to 4.0]
  Day 14 | 0 [0 to 2.0] | 0 [0 to 4.5]
  Day 21 | 0 [0 to 3.0] | 0.5 [0 to 4.5]
  Day 28 | 0 [0 to 1.0] | 1.0 [0 to 5.0]

17. Other Pre Specified Outcome: Change in "Average" Phantom Limb Pain at 6 and 12 Months From the Baseline Measurement (as Measured With the 0-10 Numeric Rating Scale)
Description: The "average" phantom limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain. The data presented is the change in the "average" phantom limb pain at 6 and 12 months from the baseline measurement.
Time Frame: 6 and 12 months following baseline (the day of the initiation of the initial intervention)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% Only (no Placebo Crossover) | Placebo Infusion Only (no Ropivacaine 0.5% Crossover) | Ropivacaine 0.5% Followed by Placebo Infusion | Placebo Followed by Ropivacaine 0.5% Infusion
Number analyzed (Participants) | 46 | 33 | 25 | 40
score on a scale
  6 month | -3.0 [-5.0 to 0] | -1.5 [-5.0 to 0] | 0 [-1.8 to 1.0] | -1.5 [-3.5 to 0]
  12 month | -2.5 [-4.0 to -0.5] | -2.0 [-5.0 to 0] | -1.0 [-4.0 to 0] | -1.0 [-3.0 to 0]

18. Other Pre Specified Outcome: Change in "Worst" Phantom Limb Pain at 6 and 12 Months From the Baseline Measurement (as Measured With the 0-10 Numeric Rating Scale)
Description: The "worst" phantom limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain. The data presented is the change in the "worst" phantom limb pain at 6 and 12 months from the baseline measurement.
Time Frame: 6 and 12 months following baseline (the day of the initiation of the initial intervention)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% Only (no Placebo Crossover) | Placebo Infusion Only (no Ropivacaine 0.5% Crossover) | Ropivacaine 0.5% Followed by Placebo Infusion | Placebo Followed by Ropivacaine 0.5% Infusion
Number analyzed (Participants) | 46 | 33 | 25 | 40
score on a scale
  6 months | -2.0 [-6.0 to 0] | -2.5 [-5.0 to 0] | 0 [-2.0 to 1.0] | -1.0 [-3.0 to 0]
  12 months | -2.0 [-4.0 to 0] | -1.0 [-5.0 to 0] | 0 [-2.0 to 1.0] | -1.5 [-3.3 to 0]

19. Other Pre Specified Outcome: Change in "Average" Residual Limb Pain at 6 and 12 Months From the Baseline Measurement (as Measured With the 0-10 Numeric Rating Scale)
Description: The "average" residual limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain. The data presented is the change in the "average" residual limb pain at 6 and 12 months from the baseline measurement.
Time Frame: 6 and 12 months following baseline (the day of the initiation of the initial intervention)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% Only (no Placebo Crossover) | Placebo Infusion Only (no Ropivacaine 0.5% Crossover) | Ropivacaine 0.5% Followed by Placebo Infusion | Placebo Followed by Ropivacaine 0.5% Infusion
Number analyzed (Participants) | 46 | 33 | 25 | 40
score on a scale
  6 months | -1.0 [-3.0 to 0] | 0 [-2.0 to 0] | 0 [-0.25 to 0] | -1.0 [-2.0 to 0]
  12 months | -2.0 [-4.0 to 0] | 0 [-3.5 to 0] | 0 [-2.0 to 0] | -1.0 [-1.5 to 0]

20. Other Pre Specified Outcome: Change in "Worst" Residual Limb Pain at 6 and 12 Months From the Baseline Measurement (as Measured With the 0-10 Numeric Rating Scale)
Description: The "worst" residual limb pain experienced over the previous 3 days evaluated with the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain. The data presented is the change in the "worst" residual limb pain at 6 and 12 months from the baseline measurement.
Time Frame: 6 and 12 months following baseline (the day of the initiation of the initial intervention)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.5% Only (no Placebo Crossover) | Placebo Infusion Only (no Ropivacaine 0.5% Crossover) | Ropivacaine 0.5% Followed by Placebo Infusion | Placebo Followed by Ropivacaine 0.5% Infusion
Number analyzed (Participants) | 46 | 33 | 25 | 40
score on a scale
  6 months | -1.0 [-5.0 to 0] | 0 [-4.0 to 0] | 0 [-5.0 to 0] | 0 [-2.0 to 1.0]
  12 months | -3.0 [-7.0 to 0] | 0 [-1.0 to 0] | 0 [-1.0 to 0] | 0 [-2.0 to 1.0]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Ropivacaine 0.5%: Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of study fluid from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. This group includes subjects who received the ropivacaine infusion either as the initial treatment or crossover treatment.
- Normal Saline (Salt Water) Infusion: Electronic, programmable, portable infusion pumps will be used to administer perineural study solution at fixed rates for over 6 days. Subjects will receive a total of 1,100 mL of normal saline placebo fluid from either one (upper extremity) or two (lower extremity) pump and external reservoir combinations. The continuous basal infusion rate will be determined by catheter location: femoral 2.5 mL/h; popliteal-sciatic 5 mL/h; and infraclavicular 7.5 mL/h (37.5 mg/h for both upper and lower extremity subjects). No patient-controlled bolus dose will be included. This group includes subjects who received the saline infusion either as the initial treatment or crossover treatment.
Arm/Group | Ropivacaine 0.5% | Normal Saline (Salt Water) Infusion
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/111 | 1/98
Other Adverse Events (participants affected / at risk) | 4/111 | 4/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine 0.5% (N=111) | Normal Saline (Salt Water) Infusion (N=98)
Increased Phantom pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — A patient had increased pain Day 2 after returning home to a different state. A local hospital physician withdrew both catheters and the pain resolved. 5 months later a retained piece of the catheter was removed. His infection healed with antibiotics
OTHER ADVERSE EVENTS (reported when occurring in more than 2.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine 0.5% (N=111) | Normal Saline (Salt Water) Infusion (N=98)
Signs of possible localized infection at catheter sites (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) — 8 catheter sites showed signs of possible local infection out of 382 total catheters. All symptoms resolved within 2 days after catheter removal..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT01824082/Prot_SAP_000.pdf